CLINICAL TRIAL: NCT01747421
Title: Validation of a High-risk Versus Low-risk Referral Model in Suspected Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christian Backer Mogensen, assistant professor, University of Southern Denmark
Other Study IDs: SLB-ED-04-2012
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In Emergency Departments patients admitted with chest pain may suffer from non-significant to lifethreatening conditions.

The aim of the present study is to develop and validate a referral model in chest pain patients which divide the patients with non- significant ECG changes into high risk and low risk groups for acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* more than 15 years old

Exclusion Criteria:

* Patients with ST-elevations in ECG

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all acute admission to Emergency Department with the complaint Chestpain
Sampling Method: Non-Probability Sample
Enrollment: 495 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Acute Myocardial Infarction | 24 hours after admission

SECONDARY OUTCOMES:
cardiac event | 1 year after admission

CONTACTS AND LOCATIONS:
Locations (1):
- Kolding Hospital, Kolding, Denmark